CLINICAL TRIAL: NCT05413122
Title: Evaluating Smoking Cessation Interventions for PWH in South Africa: Efficacy, Implementation, and Cost-effectiveness
Brief Title: Evaluating Smoking Cessation Interventions for PWH in South Africa
Acronym: Tlogela
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Colorado State University (Other); New York University (Other); Perinatal HIV Research Unit of the University of the Witswatersrand (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB00335707; 1U01CA261626-01 (NIH)
Record Dates: First submitted 2022-06-03; First posted 2022-06-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation; HIV; Comorbidities and Coexisting Conditions
Keywords: Smoking Cessation; Combination NRT; Varenicline; Behavioral Counselling; Peer Counseling
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine Chewing Gum; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a 4-factor, balanced full factorial randomized controlled trial to evaluate the main and interaction effects of these 2-level interventions in one peri-urban and one urban setting in South Africa. The investigators will randomize adults with HIV who are current smokers into 1 of 16 possible combinations of the four intervention components.
Masking Description: This will be an open-label trial; neither the participants nor study personnel will be blinded to treatment assignment post randomization, but randomization block assignment will be concealed from the study personnel who will be enrolling participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Intensive Behavioral Counselling (Experimental): Participants randomized to the Intensive Behavioural Counselling condition will receive in-person intensive (~45 minutes) behavioural counselling in the clinic at screening and at weeks 2, 4, 8, and 12. Additionally, on non-clinic visit weeks participants will receive (1) one phone call each week from the clinic counsellor, and (2) two text messages each week providing encouragement and advice. ].
  Interventions: Behavioral: Intensive Behavioral Counselling
- Peer Support (Experimental): Participants randomized to receive Peer Support will be engaged by participants' own peer counsellor over weeks -2 to 12. Peer counselling will follow a flexible framework for contact with participants, which will include in-person and phone-based check-ins, depending upon individual participant preference. Peer counsellors will visit the counsellors' assigned participant in-person at participants' home, workplace, or other setting based on participant preference at least during weeks -2, 2, 4, 8 and 12; additional in-person contact will be provided upon participant request.
  Interventions: Behavioral: Peer Counselling
- c-NRT (Experimental): A 12-week course of nicotine patches and nicotine gum will be dispensed to the participant by the counsellor according to randomization into the c-NRT condition. c-NRT will be provided per label instructions given number of cigarettes the participant smokes per day and will be provided in the commercially available package. Participants will be provided with education on its use, including where and how to place a patch, strength of patches to use and how to taper, not smoking while using the patch, and using gum ad hoc; the investigators will also discuss possible side effects. Participants will be given a number to call should the participants require assistance, and weekly calls will be made to participants to screen for adverse events and monitor adherence; calls will taper to every other week after four weeks.
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum
- Varenicline (Experimental): At enrolment, a 12-week course of varenicline in the commercially available package will be dispensed by a study clinician according to randomization into the varenicline condition and participants will be provided with education on its use. Participants will be instructed to begin taking varenicline one week prior to participants' quit date and for 11 weeks following quit date. Participants will be given a number to call should the participants require assistance, and weekly calls will be made to participants to screen for adverse events and to monitor adherence; calls will taper to every other week after four weeks.
  Interventions: Drug: Varenicline
- Control (No Intervention): No intervention
- Varenicline & c-NRT (Experimental): Varenicline & c-NRT
  Interventions: Drug: Varenicline; Drug: Nicotine patch; Drug: Nicotine gum
- Peer Support & Varenicline (Experimental): Peer Support & Varenicline
  Interventions: Drug: Varenicline; Behavioral: Peer Counselling
- c-NRT & Peer Support (Experimental): c-NRT & Peer Support
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Peer Counselling
- c-NRT & Peer Support & Varenicline (Experimental): c-NRT & Peer Support & Varenicline
  Interventions: Drug: Varenicline; Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Peer Counselling
- Intensive Behavioral Counseling & Varenicline (Experimental): Intensive Behavioral Counseling & Varenicline
  Interventions: Drug: Varenicline; Behavioral: Intensive Behavioral Counselling
- Intensive Behavioral Counseling & c-NRT (Experimental): Intensive Behavioral Counseling & c-NRT
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Intensive Behavioral Counselling
- Intensive Behavioral Counseling & Varenicline & c-NRT (Experimental): Intensive Behavioral Counseling & Varenicline & c-NRT
  Interventions: Drug: Varenicline; Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Intensive Behavioral Counselling
- Intensive Behavioral Counseling & Peer Support (Experimental): Intensive Behavioral Counseling & Peer Support
  Interventions: Behavioral: Intensive Behavioral Counselling; Behavioral: Peer Counselling
- Intensive Behavioral Counseling & Peer Support & Varenicline (Experimental): Intensive Behavioral Counseling & Peer Support & Varenicline
  Interventions: Drug: Varenicline; Behavioral: Intensive Behavioral Counselling; Behavioral: Peer Counselling
- Intensive Behavioral Counseling & Peer Support & c-NRT (Experimental): Intensive Behavioral Counseling & Peer Support & c-NRT
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Intensive Behavioral Counselling; Behavioral: Peer Counselling
- Intensive Behavioral Counseling & Peer Support & c-NRT & Varenicline (Experimental): Intensive Behavioral Counseling & Peer Support & c-NRT & Varenicline
  Interventions: Drug: Varenicline; Drug: Nicotine patch; Drug: Nicotine gum; Behavioral: Intensive Behavioral Counselling; Behavioral: Peer Counselling

INTERVENTIONS:
Drug: Varenicline — At enrolment, a 12-week course of varenicline in the commercially available package will be dispensed by a study clinician.
  Arms: Intensive Behavioral Counseling & Peer Support & Varenicline; Intensive Behavioral Counseling & Peer Support & c-NRT & Varenicline; Intensive Behavioral Counseling & Varenicline; Intensive Behavioral Counseling & Varenicline & c-NRT; Peer Support & Varenicline; Varenicline; Varenicline & c-NRT; c-NRT & Peer Support & Varenicline
Drug: Nicotine patch — A 12-week course of nicotine patches and nicotine gum will be dispensed to the participant by the counsellor according to randomization into the c-NRT condition. c-NRT will be provided per label instructions given number of cigarettes the participant smokes per day and will be provided in the commercially available package.
  Other Names: combination nicotine replacement therapy
  Arms: Intensive Behavioral Counseling & Peer Support & c-NRT; Intensive Behavioral Counseling & Peer Support & c-NRT & Varenicline; Intensive Behavioral Counseling & Varenicline & c-NRT; Intensive Behavioral Counseling & c-NRT; Varenicline & c-NRT; c-NRT; c-NRT & Peer Support; c-NRT & Peer Support & Varenicline
Drug: Nicotine gum — A 12-week course of nicotine patches and nicotine gum will be dispensed to the participant by the counsellor according to randomization into the c-NRT condition. c-NRT will be provided per label instructions given number of cigarettes the participant smokes per day and will be provided in the commercially available package.
  Other Names: nicotine replacement
  Arms: Intensive Behavioral Counseling & Peer Support & c-NRT; Intensive Behavioral Counseling & Peer Support & c-NRT & Varenicline; Intensive Behavioral Counseling & Varenicline & c-NRT; Intensive Behavioral Counseling & c-NRT; Varenicline & c-NRT; c-NRT; c-NRT & Peer Support; c-NRT & Peer Support & Varenicline
Behavioral: Intensive Behavioral Counselling — Participants randomized to the Intensive Behavioural Counselling condition will receive in-person intensive (~45 minutes) behavioural counselling in the clinic at screening and at weeks 2, 4, 8, and 12. Additionally, on non-clinic visit weeks participants will receive (1) one phone call each week from the clinic counsellor, and (2) two text messages each week providing encouragement and advice.
  Arms: Intensive Behavioral Counseling & Peer Support; Intensive Behavioral Counseling & Peer Support & Varenicline; Intensive Behavioral Counseling & Peer Support & c-NRT; Intensive Behavioral Counseling & Peer Support & c-NRT & Varenicline; Intensive Behavioral Counseling & Varenicline; Intensive Behavioral Counseling & Varenicline & c-NRT; Intensive Behavioral Counseling & c-NRT; Intensive Behavioral Counselling
Behavioral: Peer Counselling — Participants randomized to the Peer Support condition will be engaged by a peer counsellor over weeks -2 to 12. Peer counselling will follow a flexible framework for contact with participants, which will include in-person and phone-based check-ins, depending upon individual participant preference. Peer counsellors will visit the counsellors' assigned participant in-person at participants' home, workplace, or other setting based on participant preference at least during weeks -2, 2, 4, 8 and 12; additional in-person contact will be provided upon participant request.
  Other Names: Peer Support
  Arms: Intensive Behavioral Counseling & Peer Support; Intensive Behavioral Counseling & Peer Support & Varenicline; Intensive Behavioral Counseling & Peer Support & c-NRT; Intensive Behavioral Counseling & Peer Support & c-NRT & Varenicline; Peer Support; Peer Support & Varenicline; c-NRT & Peer Support; c-NRT & Peer Support & Varenicline

SUMMARY:
The overall objective of the study is to optimize a smoking cessation treatment package for people with HIV (PWH) that can be integrated into existing HIV care in South Africa.

DETAILED DESCRIPTION:
This project will evaluate the main and interaction effects of four evidence-based smoking cessation components integrated within HIV care in South Africa: (1) intensive behavioural counselling, (2) peer support, (3) combination nicotine replacement therapy (c-NRT), and (4) varenicline. The investigators will also evaluate the implementation and cost-effectiveness of these interventions. This study is a balanced full factorial randomised trial of 660 adults with HIV and will be implemented in two diverse sites in Gauteng, South Africa representing both peri-urban and urban settings.

Participants will be recruited via health care worker-referral or self-referral. Interested patients will be further screened for eligibility. Eligible participants will be administered written informed consent (see "Informed Consent and Assent" section below), and participants will be randomized into one of 16 study conditions for a 12-week intervention period. This will be an open-label trial; neither the participants nor study personnel will be blinded to treatment assignment post randomization, but randomization block assignment will be concealed from the study personnel who will be enrolling participants.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age, and
2. attend one of the selected study clinics, and
3. have a confirmed diagnosis of HIV (evidenced by one of: clinic or hospital prescription for combination antiretroviral therapy (ART), or a current ART medication pack that has the patient's name documented thereon) and
4. have been taking ART for at least three consecutive months (to ensure engagement in care at the recruitment clinic), and
5. are current tobacco smokers (smoked at least 100 cigarettes in the subject's lifetime, have smoked daily for the past 30 days, have exhaled breath carbon monoxide (CO) ≥ 7 parts per million (ppm), and have a positive urine cotinine test), and
6. either own or have household access to a mobile phone, and
7. provide written informed consent.

Exclusion Criteria:

1. Currently (within the previous 14 days) receiving or using smoking cessation counselling or pharmacotherapy, or
2. are unable to participate due to severity of medical illness, guided by a Karnofsky score of ≤ 40, or
3. have a history of seizures, cancer, heart disease, stroke, myocardial infarction, stomach ulcers, kidney failure, or liver failure, or
4. have generalized eczema or psoriasis, or
5. have cognitive dysfunction or psychosis as defined by the Mini-International Neuropsychiatric Interview (M.I.N.I.), or
6. have suicide risk as defined by the Columbia-Suicide Severity Rating Scale (C-SSRS), or
7. are pregnant, planning to become pregnant in the next four months, lactating, or are unwilling to use effective birth control, or
8. have a history of adverse reactions to varenicline or nicotine patch, or
9. are not planning to continue to receive care at the clinic for the next 52 weeks.
10. In the opinion of the attending investigator are not a candidate for the clinical trail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence tobacco abstinence at 52 weeks | 52 weeks
  Verified by exhaled breath CO < 7ppm and a negative urine cotinine test.

SECONDARY OUTCOMES:
7-day point prevalence tobacco abstinence at 26 weeks | 26 weeks
  Verified by exhaled breath CO < 7ppm and a negative urine cotinine test. Urine cotinine will be excluded as an indicator of abstinence for those self-reporting c-NRT use in the preceding week.
7-day point prevalence tobacco abstinence at 12 weeks | 12 weeks
  Verified by exhaled breath CO < 7ppm and a negative urine cotinine test. Urine cotinine will be excluded as an indicator of abstinence for those self-reporting c-NRT use in the preceding week.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Martison, Principal Investigator — Perinatal HIV Research Unit (PHRU); Jonathan E Golub, PhD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Perinatal HIV Research Unit (PHRU), Soweto, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Intellectual property and data generated under this project will be administered in accordance with policies of the Johns Hopkins University, the Perinatal HIV Research Unit (PHRU) at the University of the Witwatersrand, and NIH policies, including the most recent NIH Data Sharing Policy and Implementation Guidance. Materials generated under the project will be disseminated in accordance with University/Participating institutional and NIH policies.
  Access to data generated under the project will be available for educational, research and non-profit purposes. Publication of data shall occur during the project, as appropriate, or at the end of the project, consistent with normal scientific practices. Research data which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for sharing following publication of primary findings from the study, indefinitely.
Access Criteria: Following publication of research findings, the final research database may be shared upon request with qualified individuals within the scientific community for research purposes in accordance with the policies of the partnering organizations. Data will be stripped of all personal identifiers and available as a tab delimited ASCII data file with an accompanying data dictionary. Data will be anonymized and maintained in a password-protected database.

REFERENCES:
- [Derived] Genade LP, Steiner L, Nabeemeeah F, Niaura RS, Nonyane BAS, Hoffmann CJ, Sohn H, Kemp CG, Guastaferro K, Mlambo L, Chetty D, Waja Z, Martinson N, Golub JE, Elf JL. Evaluating smoking cessation interventions for people living with HIV in a factorial randomised clinical trial in South Africa using the Multiphase Optimization Strategy (MOST) framework: The Tlogela Trial protocol. Contemp Clin Trials. 2025 Aug;155:107985. doi: 10.1016/j.cct.2025.107985. Epub 2025 Jun 19. PMID 40543725